CLINICAL TRIAL: NCT04571957
Title: Expanding Donor Pool for Live Donor Liver Transplantation: Utilization of Donors With NASH After Optimization
Status: Completed | Type: Observational
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Other Study IDs: ILBS-LIVEDONORS-03
Record Dates: First submitted 2020-09-09; First posted 2020-10-01 (Actual); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Non Alcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Donors with NASH: Donors with NASH underwent donor optimization protocol
  Interventions: Other: No Intervention
- Donors without NASH: Donors without NASH
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No Intervention

SUMMARY:
Live donor liver transplantation (LDLT) is the treatment of choice for end-stage liver disease, predominantly in the East, where deceased donor liver transplantation is sparse. In LDLT, donor selection has to be stringent; as the donor safety is thepriority. Live liver donors (LLD) with complex biliary and vascular anatomy are increasingly being accepted for donation with the betterment of technical expertise. One of the commonest reasons for LLD rejection is the hepatic parenchymal abnormality because ofsteatosis and steatohepatitis, which can increase the donor risk. Retrospective analysis of donors with non-alcoholic steatohepatitis(NASH) who were optimized and taken up for major hepatectomy from June 2011 to January 2018will be performed.

DETAILED DESCRIPTION:
Study Design Aim and Objective -

* Primary objective:
* To study the effect of donor optimization protocol in donors with biopsy proven NASH
* To study thebiochemical (LFTSs & INR) recovery in donors with NASH after major hepatectomy
* To compare their biochemical recovery parameters (LFTs & INR) with that of non NASH donors.
* Secondary objectives:
* To study incidence of NASH among live liver donors
* To study their respective recipients' outcomes
* To study the morbidity among LLDs with NASH after major hepatectomy

Methodology:

* Study population:Patients underwentLDLT from June 2011 to January 2019 at Institute of Liver & Biliary Sciences, New Delhi
* Study design:Retrospective study
* Study period:from June 2011 to January 2019
* Sample size with justification:All consecutive LLDs with at least one year of follow up post-operatively
* Intervention: none
* Monitoring and assessment:none Statistical Analysis:Categorical variables were presented as number (percentage) and were compared using the Chi-square test. Continuous variables were presented as mean (standard deviation, SD) and were compared using Mann-Whitney U Test.

Adverse Effects: None Stopping Rule of Study: None

Expected Outcome of the Project: Adherence to a strict dietary and lifestyle modifications plan will cause histological reversal of NASH and fibrosis in LLDs. Their clinical and biochemical recovery following the major hepatectomy will be similar to that of non-NASH LLDs.

ELIGIBILITY:
Inclusion Criteria:

1. Live Liver Donors who had undergone major hepatectomy (removal of ≥ 3 liver segments)

Exclusion Criteria:

1. Live Liver Donors who had undergone minor hepatectomy (removal of < 3 liver segments)
2. Live Liver Donors of recipients with acute liver failure.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients underwent LDLT from June 2011 to January 2019 at Institute of Liver & Biliary Sciences, New Delhi
Sampling Method: Non-Probability Sample
Enrollment: 410 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Effect of donor optimization protocol on body weight in donors with biopsy proven NASH | 6 weeks to 3 months
Effect of donor optimization protocol on liver attenuation index in donor with biopsy proven NASH. | 6 weeks to 3 months
Effect of donor optimization protocol on lipid profile in donors with biopsy proven NASH. | 6 weeks to 3 months
Effect of donor optimization protocol on Liver Function Test in donors with biopsy proven NASH. | 6 weeks to 3 months
Improvement in Liver Function Test in donors with NASH after major hepatectomy. | Day 0 to Day 7
Improvement in Coagulation Profile in donors with NASH after major hepatectomy. | Day 0 to Day 7
Improvement in Liver Function Test between both the groups | Day 0 to Day 7

SECONDARY OUTCOMES:
Proportion of NASH among live liver donors | Day 0
Morbidity among Live Liver Donors with NASH after major hepatectomy | Day 0 to Day 30
Post Operative complications of recipients in both the groups | Day 0 to day 30

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided